CLINICAL TRIAL: NCT02283151
Title: The Effects of a Very Low Carbohydrate Diet Intervention on Weight Control in Overweight/Obese Patients in China
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Southern Medical University, China (Other)
Responsible Party: Principal Investigator, Jia Sun, Attending Doctor, Southern Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Grant No.81300689
Record Dates: First submitted 2014-10-26; First posted 2014-11-05 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-10

CONDITIONS: Overweight
Keywords: Very Low Carbohydrate Diet; Overweight/obese
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- energy-restricted diet (Other): The control group was given an energy-restricted diet (ER diet). Energy-restricted diet was designed in the traditional Chinese style with an initial target for a total energy intake of 1200 kcal/d (5021 kJ/d). Supplementation of multivitamins and minerals was provided per day.
  Interventions: Other: energy-restricted diet
- diet nutrition bar (Experimental): The experimental group was given individual instructions on how to follow the VLCD (very low carbohydrate diet). Energy intake was restricted to less than 800kcal/day (3349kJ/d) (carbohydrate intake < 20g/d). Carbohydrate-rich foods, such as white rice, steamed bread and tubers, were substituted with fish, poultry and plant oil. All daily meals were replaced as follows: a cup of soybean milk (200 mL) and a boiled egg at breakfast; a diet nutrition bar (106 Kcal: 2.8 g carbohydrate, 11.2 g protein and 5.6 g fat; Nutriease Health Technology Co., Ltd., Hangzhou, China), nonstarchy vegetables (<200 kcal), and 50 g protein from meat (i.e., beef, lean pork, skinned chicken, fish) at lunch and dinner. Supplementation of multivitamins and minerals was provided per day.
  Interventions: Dietary Supplement: diet nutrition bar

INTERVENTIONS:
Dietary Supplement: diet nutrition bar — The experimental group was given individual instructions on how to follow the VLCD (very low carbohydrate diet). Energy intake was restricted to less than 800kcal/day (3349kJ/d) (carbohydrate intake < 20g/d). All daily meals were replaced as follows: a cup of soybean milk (200 mL) and a boiled egg at breakfast; a diet nutrition bar(Nutriease Health Technology Co., Ltd., Hangzhou, China), nonstarchy vegetables (<200 kcal), and 50 g protein from meat at lunch and dinner. Supplementation of multivitamins and minerals was provided per day.
  Arms: diet nutrition bar
Other: energy-restricted diet — The control group was given an energy-restricted diet (ER diet). Energy-restricted diet was designed in the traditional Chinese style with an initial target for a total energy intake of 1200 kcal/d (5021 kJ/d).
  Arms: energy-restricted diet

SUMMARY:
The study was designed to investigate the effects of a very low carbohydrate diet (VLCD) intervention on weight control in overweight/obese patients in China.All the subjects were randomly assigned to experiment group and control group. The experimental group was given individual instructions on how to follow the VLCD (very low carbohydrate diet). The control group was given an energy-restricted diet.The energy-restricted diet (ER diet) was designed in the traditional Chinese style with an initial target for a total energy intake of 1200 kcal/d (5021 kJ/d).

DETAILED DESCRIPTION:
121 obese or overweight patients were enrolled in the study and 23 patients were dropped out (43 male, 55 female, aged≥18 years, BMI≥24 kg/m2) from the outpatient clinic of endocrinology and metabolism department of Southern Medical University Affiliated ZhuJiang Hospital. All the subjects were randomly assigned to experiment group and control group. The experimental group was given individual instructions on how to follow the VLCD (very low carbohydrate diet). Energy intake was restricted to less than 800kcal/day (3349kJ/d) (carbohydrate intake < 20g/d). All daily meals were replaced as follows: a cup of soybean milk (200 mL) and a boiled egg at breakfast; a diet nutrition bar (106 Kcal: 2.8 g carbohydrate, 11.2 g protein and 5.6 g fat; Nutriease Health Technology Co., Ltd., Hangzhou, China), nonstarchy vegetables (<200 kcal), and 50 g protein from meat (i.e., beef, lean pork, skinned chicken, fish) at lunch and dinner. Supplementation of multivitamins and minerals was provided per day. The energy-restricted diet (ER diet) was designed in the traditional Chinese style with an initial target for a total energy intake of 1200 kcal/d (5021 kJ/d). Subjects were also encouraged to drink at least 1.8 litres of water per day, and asked to maintain their habitual level of physical activity. Compliance with the diet and physical activity level was checked at weekly visits.

ELIGIBILITY:
Inclusion Criteria:

* overweight or obese healthy volunteers (43 male, 55 female, aged≥18years, BMI≥24 kg/m2)

Exclusion Criteria:

* pregnant or plan for pregnant
* lactation or postmenopausal women
* use of any prescription medication in previous 2 months
* had any weight loss diet or pill during the past 6 months
* consuming>20 g/day of alcohol
* tobacco use within 6 month
* cardiovascular or endocrine disease history
* hypertension history or current elevated blood pressure (systolic blood pressure (SBP): ≥150 mmHg; diastolic blood pressure (DBP)≥90 mmHg; current treatment for hypertension)
* diabetes mellitus
* acute or chronic infections
* hepatopathy, kidney disease, gastrointestinal disease or any other acute or chronic diseases requiring treatment.

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2013-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
body composition | before intervention and after 12 weeks' intervention
  body composition included weight, body mass index, body fat, body fat percentage, visceral fat, waist-to-hip ratio

CONTACTS AND LOCATIONS:
Overall Officials: Jia Sun, PhD., Principal Investigator — Southern Medical University, China